CLINICAL TRIAL: NCT02038296
Title: Different Protocols for Repeated Transarterial Chemoembolization in the Treatment of Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: TAE001
Record Dates: First submitted 2014-01-15; First posted 2014-01-16 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Liver Cancer
Keywords: Hepatocellular carcinoma; Transarterial chemoembolization; Gemcitabine
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Group 1 (Experimental): Group 1 received single-drug (doxorubicin)transarterial chemoembolization.
  Interventions: Procedure: transarterial chemoembolization
- Group 2 (Experimental): Group 2 received double-drug (doxorubicin and mitomycin C)transarterial chemoembolization
  Interventions: Procedure: transarterial chemoembolization
- Group 3 (Experimental): Group 3 were treated with triple-drug (doxorubicin, mitomycin C and gemcitabine)transarterial chemoembolization.
  Interventions: Procedure: transarterial chemoembolization

INTERVENTIONS:
Procedure: transarterial chemoembolization

SUMMARY:
To evaluate local tumor control and survival rate after repeated transarterial chemoembolization(TACE) using three different protocols in hepatocellular carcinoma (HCC) patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed HCC with unresectable disease without extrahepatic metastases;
* HCC with no previous treatment;
* age between 18 and 75 years;
* Life expectancy of at least 8 weeks;
* main tumor size greater than 5 cm;
* adequate hematologic function (platelet count: >60 × 109 platelets/L; hemoglobin: >90g/L; and prothrombin time: <3 seconds above control);
* adequate renal function (serum creatinine: ≤1.5 × upper limit of normal);
* Child-Pugh classification A or B grade;
* Barcelona Clinic Liver Cancer (BCLC) stage B or C;
* Eastern Co-operative Group performance status of zero or one.

Exclusion Criteria:

* a hypovascular tumor (defined as a tumor with all its parts less contrast-enhanced than the nontumorous liver parenchyma on arterial phase computed tomography scans);
* diffuse-type HCC;
* evidence of hepatic decompensation including esophageal or gastric variceal bleeding or hepatic encephalopathy;
* severe underlying cardiac or renal diseases;
* color Doppler ultrasonography showing portal vein tumor thrombosis with complete main portal vein obstruction without cavernous transformation; or obstructive jaundice.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2008-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
overall survival | 1-2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Interventional Radiology; Cancer Center; Guangdong General Hospital, Guangzhou, Guangdong, China